CLINICAL TRIAL: NCT06794372
Title: [68Ga]Ga-FAPI-46 PET/CT in Early Detection of Lymph Node Metastasis in Head and Neck Squamous Cell Carcinomas
Brief Title: [68Ga]Ga-FAPI-46 in Staging of Head and Neck Carcinomas
Acronym: FAPIHN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: John O. Prior (Other)
Responsible Party: Sponsor-Investigator, John O. Prior, MD, PhD, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPIHN; 2024-01881 (Registry Identifier: BASEC)
Record Dates: First submitted 2024-12-24; First posted 2025-01-27 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma HNSCC
Keywords: Head and Neck Squamous Cell Carcinoma; Cancer-associated fibroblasts; PET/CT; Lymph nodes; Tumor microenvironment; Fibroblast activation protein
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HNSCC patients (Experimental): Patients with operable head and neck cancer presenting histologically proven HNSCC, planned to undergo surgery (tumour and lymph node dissection), and who will benefit, as standard of care, from cervical MRI, ceCT and 18F-FDG PET/CT.
  Interventions: Drug: [68Ga]Ga-FAPI-46 PET/CT

INTERVENTIONS:
Drug: [68Ga]Ga-FAPI-46 PET/CT — [68Ga]Ga-FAPI-46 PET/CT

SUMMARY:
The trial focuses on assessing the role of [68Ga]Ga-FAPI-46 in head and neck squamous cell carcinomas (HNSCC) staging before surgery. In the context of metastasis, cancer-associated fibroblasts (CAFs) emerge as pivotal contributors to the creation of a microenvironment conducive to future metastases. CAFs exert their influence through intricate mechanisms, including the remodeling of the extracellular matrix by secreting proteins such as collagen and fibronectin. This process enhances the structural support for cancer cell invasion into adjacent tissues. Additionally, CAFs play a central role in promoting angiogenesis, ensuring an adequate blood supply to the tumor, which may also facilitate the entry of cancer cells into the bloodstream. Through modulation of immune responses within the tumor microenvironment, CAFs establish an immunosuppressive milieu, providing a permissive environment for cancer cell survival and dissemination. Collectively, the orchestrated activities of CAFs contribute to the preparation of a metastatic niche, influencing the microenvironment at both primary and secondary sites and enhancing the likelihood of successful metastasis.

Employing [68Ga]Ga-FAPI-46 PET/CT imaging to target activated CAFs may hold the potential to discern lymph nodes (LNs) predisposed to future metastases in HNSCC. The use of this imaging modality offers a unique opportunity to visualize and assess the presence and activity of CAFs within the tumor microenvironment. By targeting the fibroblast activation protein (FAP), a receptor enriched on CAFs, this imaging approach provides a specific and sensitive mean to identify regions where the microenvironment may favor metastatic progression.

In this research endeavor, the primary objective is to highlight the additional value of [68Ga]Ga-FAPI-46 PET/CT into the standard pre-surgical imaging protocol. Additionally, the study will evaluate the efficacy of FAP positon emission tomography (PET) in primary tumor delineation. Imaging based on [68Ga]Ga-FAPI-46 allows the identification of CAFs, specifically by exploiting their increased FAP expression. The study aims also to systematically compare the [68Ga]Ga-FAPI-46 PET/CT signals with the characteristics of resected lymph nodes, seeking to ascertain the capability of FAPI PET imaging in identifying premetastatic conditions. By comparing the [68Ga]Ga-FAPI-46 PET signal and the histopathological features of resected lymph nodes, the goal is to validate the potential of [68Ga]Ga-FAPI-46 PET imaging as a tool for early detection of premalignant or metastatic conditions in the lymphatic system before surgical intervention. The ability to pinpoint lymph nodes at risk for future metastases could revolutionize clinical decision-making, by facilitating a more nuanced understanding of disease spread, thereby informing personalized treatment strategies and potentially improving patient outcomes.

DETAILED DESCRIPTION:
[68Ga]Ga-FAPI-46 PET/CT is an advanced imaging technique utilized in nuclear medicine for the evaluation of various cancers. The imaging agent [68Ga]Ga-FAPI-46 specifically targets FAP, a protein overexpressed by CAFs in the tumor microenvironment. This targeted approach allows for precise visualization of FAP-positive tumors, aiding in the detection, staging, and assessment of therapeutic response. The integration of PET and CT modalities provides both functional and anatomical information, enhancing the accuracy of the imaging results. In this study, the investigators will specifically evaluate the application of [68Ga]Ga-FAPI-46 PET/CT in patients diagnosed with HNSCC who are scheduled for primary clinical resection. This research aims to explore the potential of [68Ga]Ga-FAPI-46 PET/CT in guiding treatment decisions and optimizing the management of HNSCC, contributing valuable insights to the growing knowledge in precision oncology.

Patients with confirmed HNSCC and planned to undergo tumor and LN dissection surgery will be recruited for this project. The included patients will follow their standard-of-care clinical investigations according to current guideline-based recommendations.

Patients will receive [68Ga]Ga-FAPI-46 in a dose of 2MBq/kg (+/-15%) as an IV injection. The total administered dose will be between 80 and 200MBq. 60 minutes (+/- 10min) after the injection, low-dose, non-contrast-enhanced PET/CT will be acquired for about 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Karnofsky index ≥80%
* Patients with operable head and neck cancer presenting histologically proven HNSCC (including Oral Cavity Cancer, Pharyngeal Cancer, Laryngeal Cancer)
* Patients with at least one nodal metastasis
* Patients scheduled for neck dissection
* SOC imaging (MRI, ceCT and 18F-FDG-PET/CT) performed as pre-surgery exams
* Written informed consent obtained

Exclusion Criteria:

* Known pregnancy or ongoing breast feeding
* Claustrophobia
* Severe renal insufficiency (GFR<30 mL/min/1,73 m2)
* Liver enzymes (ALAT, ASAT)>5 times the standard upper limit
* Bilirubin>3 times the standard upper limit
* Hemoglobin<8 g/dL
* Absolute neutrophil count<1000/mm3
* Platelets<75000/µL
* insufficient knowledge of project language, inability to give consent or to follow trial-associated procedures
* the patient makes use of his/her "right not to know" and refuses to be informed about incidental findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
[68Ga]Ga-FAPI-46 PET/CT imaging results: tumor size | 6 weeks
  The tumor size (mm*mm) measured by 68Ga-FAPI-46 PET/CT will be reported. Results will be compared to the clinically indicated standard imaging (FDG PET/CT, ceCT and MRI).
[68Ga]Ga-FAPI-46 PET/CT imaging results: tumor volume | 6 weeks
  The tumor volume (mm^3) measured by 68Ga-FAPI-46 PET/CT will be reported. Results will be compared to the clinically indicated standard imaging (FDG PET/CT).
[68Ga]Ga-FAPI-46 PET/CT imaging results: tumor SUVmax | 6 weeks
  The SUVmax of the tumor measured by 68Ga-FAPI-46 PET/CT will be reported. Results will be compared to the clinically indicated standard imaging (FDG PET/CT).
[68Ga]Ga-FAPI-46 PET/CT imaging results: number of lesions | 6 weeks
  The number of lesions (for nearby lymph nodes and distant metastases) visible by 68Ga-FAPI-46 PET/CT will be reported.
  Results will be compared to the clinically indicated standard imaging (FDG PET/CT, ceCT and MRI).
[68Ga]Ga-FAPI-46 PET/CT imaging results: lesion site | 6 weeks
  The site of lesions (for nearby lymph nodes and distant metastases) visible by 68Ga-FAPI-46 PET/CT will be reported.
  Results will be compared to the clinically indicated standard imaging (FDG PET/CT, ceCT and MRI).
[68Ga]Ga-FAPI-46 PET/CT imaging results: lesion size | 6 weeks
  The size (mm*mm) of lesions (for nearby lymph nodes and distant metastases) visible by 68Ga-FAPI-46 PET/CT will be reported.
  Results will be compared to the clinically indicated standard imaging (FDG PET/CT, ceCT and MRI).
[68Ga]Ga-FAPI-46 PET/CT imaging results: lesion volume | 6 weeks
  The volume (mm^3) of lesions (for nearby lymph nodes and distant metastases) visible by 68Ga-FAPI-46 PET/CT will be reported.
  Results will be compared to the clinically indicated standard imaging (FDG PET/CT).
[68Ga]Ga-FAPI-46 PET/CT imaging results: lesion SUVmax | 6 weeks
  The SUVmax of lesions (for nearby lymph nodes and distant metastases) visible by 68Ga-FAPI-46 PET/CT will be reported.
  Results will be compared to the clinically indicated standard imaging (FDG PET/CT).
[68Ga]Ga-FAPI-46 PET/CT imaging results: TNM tumor stage | 6 weeks
  The TNM stage calculated by 68Ga-FAPI-46 PET/CT will be reported. Results will be compared to the clinically indicated standard imaging (FDG PET/CT, ceCT and MRI).

SECONDARY OUTCOMES:
Ability of [68Ga]Ga-FAPI-46 PET/CT to visualize tumor infiltration in lymph nodes | 2 months
  Histopathology of clinically indicated resected lymph node specimen will be performed. [68Ga]Ga-FAPI-46 PET/CT results and tumor infiltration findings by histology will be compared (lesions defined positive/negative as a result of the two techniques).

OTHER OUTCOMES:
Evaluation of FAP+ CAFs distribution | 1 year
  Presence (positive/negative) of FAP+ cells in tumor center, tumor invasive margin and adjacent normal tissue.
Comparison of [68Ga]Ga-FAPI-46 PET/CT with FAP immunoistochemistry | 1 year
  The ability of [68Ga]Ga-FAPI-46 PET/CT to identify FAP+ cells in lymph node lesions will be evaluated. The measurement will compare if lesions are defined as positive/negative by FAPI PET (positive/negative) and by histology showing FAP+ CAFs in the lesion.
Evaluation of desmoplastic changes | 1 year
  Resected LNs will be analyzed by histopathology to determine the presence of desmoplastic changes. Desmoplastic changes will be expressed as the expression of specific molecular markers.
Evaluation of modifications to the current therapeutic approach (questionnaire) | Questionnaire 2 ± 1 week after surgery
  Modifications to the current therapeutic approach will be evaluated by the head and neck surgeon, who will fill out a questionnaire about the foreseen therapeutic approach with and without taking into account the results of the [68Ga]Ga-FAPI-46 PET/CT. The questionnaire will contain yes/no questions or multiple choice questions.

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus Schaefer, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre hospitalier universitaire vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No